CLINICAL TRIAL: NCT07072949
Title: The Impact of Ursodeoxycholic Acid and Probiotics on Metabolic Outcomes in Type 2 Diabetic Patients Taking Metformin: a Randomized, Double-blind Clinical Trial
Brief Title: The Impact of Ursodeoxycholic Acid and Probiotics on Metabolic Outcomes in Type 2 Diabetic Patients Taking Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Banja Luka (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRUDCAT2DM
Record Dates: First submitted 2024-07-07; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Probiotics; Dietary Supplements; Ursodeoxycholic Acid

STUDY DESIGN:
Intervention Model Description: A monocentric prospective randomized double-blind controlled study included 90 patients with T2DM on metformin therapy. Patients were randomized into three groups: a metformin group (1000 to 2000 mg daily in two doses), a metformin and probiotic group (metformin + oral probiotic 3x1 capsule), and a metformin, probiotic and UDCA group (metformin + probiotic 3x1 caps + UDCA 3x1 capsule) for four weeks. Two visits were conducted during the study - at the beginning and the end. Visits involved patient interviews, clinical data collection, anthropometric measurements, biochemical analyses and stool sample analysis for the presence of probiotic culture and UDCA.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- The Metformin Group (Other)
  Interventions: Other: Metformin Monotherapy
- The Metformin/Probiotic Group (Other)
  Interventions: Other: Metformin combined with probiotic (Normia® Jadran Galenski Laboratory) supplementation
- The Metformin/Probiotic/UDCA Group (Other)
  Interventions: Other: Triple therapy - metformin, probiotic and ursodeoxycholic acid (Bilexin®, Bosnalijek)

INTERVENTIONS:
Other: Metformin Monotherapy — Participants in this group (n = 30) received metformin alone, administered in a daily dose of 1000 to 2000 mg divided into two doses, over a period of four weeks.
  Arms: The Metformin Group
Other: Metformin combined with probiotic (Normia® Jadran Galenski Laboratory) supplementation — Participants (n = 30) received metformin (1000-2000 mg/day, divided in two doses) combined with a probiotic supplement (1 capsule three times daily) over a four-week period.
  Arms: The Metformin/Probiotic Group
Other: Triple therapy - metformin, probiotic and ursodeoxycholic acid (Bilexin®, Bosnalijek) — Participants in this group (n = 30) were treated with a combination of metformin (1000 - 2000 mg/day), a probiotic (1 capsule three times daily) and ursodeoxycholic acid (UDCA, 1 capsule (250mg) three times daily) for four weeks.
  Arms: The Metformin/Probiotic/UDCA Group

SUMMARY:
A monocentric prospective randomized double-blind controlled study included 90 patients with T2DM on metformin therapy. Patients were randomized into three groups: a metformin group (1000 to 2000 mg daily in two doses), a metformin and probiotic group (metformin + oral probiotic 3x1 capsule), and a metformin, probiotic and UDCA group (metformin + probiotic 3x1 caps + UDCA 3x1 capsule) for four weeks. Two visits were conducted during the study - at the beginning and the end. Visits involved patient interviews, clinical data collection, anthropometric measurements, biochemical analyses and stool sample analysis for the presence of probiotic culture and UDCA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 25 years
* Clinical diagnosis of type 2 diabetes mellitus (T2DM) within the past 12 months
* Body mass index (BMI) ≥ 25 kg/m²
* Stable metformin therapy (1000-2000 mg daily in divided doses)
* No use of probiotics, antibiotics, vitamins, or minerals in the past 30 days

Exclusion Criteria:

* Diagnosis of type 1 diabetes mellitus
* History or diagnosis of gastrointestinal diseases
* Chronic kidney disease
* Valvular heart disease
* Pregnancy
* Presence of any acute infection

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Change in fasting plasma glucose (FPG) from baseline to week 4 | Baseline and after 4 weeks of intervention
  Fasting plasma glucose concentration will be measured in mmol/L to assess changes in glycemic control following treatment in each group.
Change in postprandial glucose (PPG) from baseline to week 4 | Baseline and after 4 weeks of intervention
  Postprandial plasma glucose concentration will be measured 2 hours after a standardized meal to evaluate treatment efficacy.
  Unit of measure: mmol/L
Change in hemoglobin A1c (HbA1c) from baseline to week 4 | Baseline and after 4 weeks of intervention
  Glycated hemoglobin (HbA1c) will be measured to assess average blood glucose levels over the preceding 4 weeks.
  Unit of measure: Percent (%)
Percentage of participants achieving HbA1c < 7.0% at week 4 | After 4 weeks of intervention
  Proportion of participants in each group achieving HbA1c values below 7.0%, indicating improved glycemic control.
  Unit of measure: Percentage of participants (%)

SECONDARY OUTCOMES:
Change in total cholesterol from baseline to week 4 | Baseline and after 4 weeks of intervention
  Assessment of total serum cholesterol levels to evaluate lipid profile modulation in response to intervention.
  Unit of measure: mmol/L
Change in LDL cholesterol from baseline to week 4 | Baseline and after 4 weeks of intervention
  Measurement of low-density lipoprotein cholesterol to assess cardiovascular risk changes.
  Unit of measure: mmol/L
Change in HDL cholesterol from baseline to week 4 | Baseline and after 4 weeks of intervention
  Measurement of high-density lipoprotein cholesterol to evaluate potential improvement in lipid metabolism.
  Unit of measure: mmol/L
Change in triglycerides from baseline to week 4 | Baseline and after 4 weeks of intervention
  Serum triglyceride levels will be measured to observe any changes due to intervention.
  Unit of measure: mmol/L
Change in C-Reactive Protein (CRP) from baseline to week 4 | Baseline and after 4 weeks of intervention
  C-reactive protein will be quantified to assess the anti-inflammatory potential of the interventions.
  Unit of measure: mg/L

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health Institution Dom zdravlja Banja Luka, Banja Luka, Republika Srpska, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Undecided